CLINICAL TRIAL: NCT02123992
Title: A Prospective, Safety and Efficacy Cohort Study of Elevate® Apical and Posterior Prolapse Repair System Compared to Native Tissue Repair for Pelvic Organ Prolapse Repair
Brief Title: Study of the Elevate Apical and Posterior Prolapse Repair System Compared to Native Tissue Repair for Pelvic Organ Prolapse
Acronym: Harmony 522
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Astora business is closing
Sponsor: ASTORA Women's Health (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PR1206
Record Dates: First submitted 2014-04-24; First posted 2014-04-28 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Elevate Apical and Posterior (Active Comparator): The experimental arm of the study will include the implantation of the Elevate Posterior surgical mesh for the treatment of posterior vaginal prolapse
  Interventions: Device: Elevate Apical and Posterior
- Native Tissue Repair (Active Comparator): The control arm of the study will include the treatment of posterior vaginal prolapse using standard surgical sutures
  Interventions: Procedure: Native Tissue Repair for pelvic organ prolapse

INTERVENTIONS:
Device: Elevate Apical and Posterior
  Arms: Elevate Apical and Posterior
Procedure: Native Tissue Repair for pelvic organ prolapse
  Arms: Native Tissue Repair

SUMMARY:
The aim of this study is to further evaluate the safety and efficacy of the Elevate® Apical and Posterior Prolapse Repair System for repair of apical/posterior pelvic organ prolapse in a controlled, post-market cohort study.

DETAILED DESCRIPTION:
The Harmony 522 study has been terminated due to the closing of the Astora Women's Health business. No other entity will be taking responsibility for this study. The study was terminated with partial subject enrollment complete and therefore no primary or secondary data analysis can be performed. The data from this study resides in a national data base which Astora no longer has access and therefore is another reason why no data analysis can be performed. The national database is owned and managed by the American Urogynecology Society (AUGS). AUGS has access to Astora's data and will at some time in the near future publish results to physicians who are active participants in the registry. Full public disclosure of this data may not occur for a number of years and will be aggregated with data from other study sponsors.

ELIGIBILITY:
Inclusion Criteria:

Subject is female

Subject is at least 18 years of age

Subject must have documented diagnosis of posterior or posterior and apical vaginal prolapse with leading edge of pelvic organ prolapse at or beyond the hymen. At or beyond the hymen is defined as POP-Q scores of Bp ≥ 0; or Bp ≥ 0 and C ≥ -1/2 TVL (for a multi-compartment posterior prolapse that includes the apical compartment)

Subject reports a bothersome bulge they can see or feel per PFDI-20, question 3, response of 2 or higher (i.e., responses of "somewhat", "moderately", or "quite a bit")

Subject or subject's legally authorized representative is willing to provide written informed consent

Subject is willing and able to comply with the follow-up regimen

Exclusion Criteria:

Subject is pregnant or intends to become pregnant during the study

Subject has an active or chronic systemic infection including any gynecologic infection, untreated urinary tract infection (UTI) or tissue necrosis

Subject has history of pelvic organ cancer (e.g. uterine, ovarian, bladder, or cervical)

Subject has had prior or is currently undergoing radiation, laser therapy, or chemotherapy in the pelvic area

Subject has taken systemic steroids (within the last month), or immunosuppressive or immunomodulatory treatment (within the last 3 months)

Subject has systemic connective tissue disease (e.g. scleroderma, systemic lupus erythematosus (SLE), Marfan's syndrome, Ehlers Danhlos, collagenosis, polymyositis or polymyalgia rheumatica)

Subject has chronic systemic pain that includes the pelvic area or chronic focal pain that involves the pelvis

Subject has uncontrolled diabetes mellitus (DM)

Subject has a known neurologic or medical condition affecting bladder function (e.g., multiple sclerosis, spinal cord injury or stroke with residual neurologic deficit)

Subject is seeking obliterative vaginal surgery as treatment for pelvic organ prolapse (colpocleisis)

Subject is not able to conform to the modified dorsal lithotomy position

Subject is currently participating in or plans to participate in another device or drug study during this study

Subject has a known sensitivity to polypropylene

Subject has had previous prolapse repair with mesh in the target compartment

Subject is planning to undergo a concomitant repair with use of mesh in the non-target compartment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2014-04; Primary Completion 2019-04 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Surgical success or failure through composite endpoint including anatomic, subjective and re-treatment measures | 36 months
Rate of device or procedure related serious adverse events | 36 months

SECONDARY OUTCOMES:
Surgical success or failure through composite endpoint including anatomic, subjective and re-treatment measures | 36 months
Rate of repeat surgery/revision for prolapse arising from the same site/target compartment | 36 months
Changes in Quality of Life measured through the following questionaires: PFDI- 20,PFIQ-7, PISQ-12 | 36 months

OTHER OUTCOMES:
Subjects experiencing adverse events related to device or procedure | 36 months
Subjects experiencing vaginal bulge | 36 months
Subjects experiencing prolapse at or beyond the hymenal ring [Time Frame: 36 months | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Eric R Sokol, MD, Principal Investigator — Stanford University
Locations (23):
- United States (23):
  - Urological Associates of Southern Arizona, Tucson, Arizona
  - The Clark Center for Urogynecology, Newport Beach, California
  - Yale School of Medicine, New Haven, Connecticut
  - National Center for Advanced Pelvic Surgery, Washington D.C., District of Columbia
  - Women's Health Advantage, Fort Wayne, Indiana
  - Metro Urology, Woodbury, Minnesota
  - Adult & Pediatric Urology and Urogynecology, Omaha, Nebraska
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - Delaware Valley Urology, Mount Laurel, New Jersey
  - Princeton Medical Center, Princeton, New Jersey
  - The Center for Specialized Women's Health, Whippany, New Jersey
  - North Shore Women's Health Clinic, Great Neck, New York
  - Premier Medical Group, Poughkeepsie, New York
  - The Institute for Female Pelvic Medicine - St. Luke's Hospital, Allentown, Pennsylvania
  - Center for Women's Health of Lansdale, Lansdale, Pennsylvania
  - The Female Pelvic Health Center, Newtown, Pennsylvania
  - Swan Urogynecology, Nashville, Tennessee
  - The Womens Centre, Denton, Texas
  - University of Texas at Galveston, Galveston, Texas
  - Lone Star Urogynecology and Continence Center, Round Rock, Texas
  - Female Pelvic Medicine Institute of Virginia, North Chesterfield, Virginia
  - Athena Women's Health, Issaquah, Washington
  - University of Washington Pelvic Health Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared at a later data by the American Urogynecology Society aggregated with other data extracted from a national registry database.